CLINICAL TRIAL: NCT00004699
Title: Dose Ranging Study of Recombinant Human Insulin-like Growth Factor I in Children With Hyperinsulinism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13381; CHP-FDR001181-DR
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-03

CONDITIONS: Hyperinsulinism
Keywords: endocrine disorders; hyperinsulinism; rare disease
MeSH Terms: conditions — Hyperinsulinism; Endocrine System Diseases; Rare Diseases | interventions — Insulin-Like Growth Factor I

INTERVENTIONS:
Drug: insulin-like growth factor I

SUMMARY:
OBJECTIVES:

I. Determine the dose of recombinant human insulin-like growth factor I that minimizes or decreases the need for exogenous glucose support without causing hypoglycemia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a dose escalation study. Patients receive an escalating dose of recombinant human insulin-like growth factor I (IGF-I). IGF-I is given subcutaneously twice a day. The dose of IGF-I is increased each day for 4 days. Glucose is administered intravenously, when necessary, to prevent hypoglycemia.

Following the study treatment patients resume prior medication and may undergo surgery.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of hyperinsulinism (i.e., evidence of fasting hypoglycemia with inadequate suppression of insulin, normal pituitary and adrenal function, and increased insulin action)
* Intractable hypoglycemia (i.e., persistent IV glucose requirement for maintaining glucose levels greater than 60 mg/dL)
* Failed standard treatment regimen of diazoxide, octreotide, and frequent feedings to control hypoglycemia
* No other major medical problems

Ages: 3 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8
Dates: Start 1995-08; Study Completion 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Pinchas Cohen, Study Chair — Children's Hospital of Philadelphia